CLINICAL TRIAL: NCT00677001
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of R306465 in Subjects With Advanced Solid Malignancies
Brief Title: A Research Study to Evaluate the Safety of R306465, a Drug in Development for Cancer and to Study the Absorption, Break Down and Elimination in Patients With Advanced Solid Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen-Cilag Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010630
Record Dates: First submitted 2008-04-24; First posted 2008-05-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Neoplasms
Keywords: Solid tumors; solid malignancies; neoplasms; refractory solid tumors; advanced solid tumors
MeSH Terms: conditions — Neoplasms | interventions — R 306465

INTERVENTIONS:
Drug: R306465

SUMMARY:
The purpose of this study is to assess the safety of R306465 (a drug in development for cancer) in patients with advanced cancer on the maximum dose that can be tolerated. Also, the absorption, breakdown and elimination of the drug will be studied.

DETAILED DESCRIPTION:
R306465, a histone deacetylase (HDAC) inhibitor, is a new drug in development for cancer. In this study, the safety (the effect on the body) of R306465 in patients with advanced cancer will be studied and the maximum dose that can be tolerated by these patients will be determined. The absorption, break down, and elimination of the drug will be studied. Antitumor activity of R306465 will be evaluated.

R306465 will be administered in a continuous regimen for 21 days followed by a 1-week rest period, which constitutes a 28-day treatment cycle. The dose of R306465 will start low and will be increased during the study in groups of 3 to 6 patients. If a group of patients does not have severe side effects, the next group of patients will get a higher dose. The dose will increase until some patients have severe side effects. The dose will then be decreased to a dose level where severe side effects are observed in less than 1/3 of patients. The amount of R306465 in the blood will be measured and the effect on the disease will be evaluated in all patients.

Patients will be screened for eligibility within 4 weeks before study treatment is given. The duration of treatment will depend on adverse effects and whether there is benefit from the treatment.

The design of a cycle may be adjusted during the course of the study as guided by clinical observations. The dosing regimen may be adjusted as guided by information on how rapidly your body breaks down and eliminates the study drug. Patients will be informed if there are changes in the design of a cycle or the dosing regimen.

During the first treatment cycle, patients are required to stay in the hospital for at least 3 nights. In addition there are 6 daytime visits during Cycles 1 and 2 (combined) that may take up to 4 hours after the morning dose. From Cycle 3 onwards, there are only 2 daytime visits per treatment cycle, and these visits usually take up less time.

Throughout the study, especially during Cycles 1 and 2, patients will undergo frequent blood and urine tests, procedures to assess safety including heart function, and tests to assess the course of the patient's illness. Two weeks after the last dose of the study drug, patients are required to return to the study site for follow-up assessments. R306465 will be administered orally once daily for 21 consecutive days followed by a 1-week rest period. These 4 weeks will constitute 1 treatment cycle. The starting dose level will be 100mg. The dose for each patient will be assigned at enrollment. On the basis of assessment by the investigator, the patient may continue to receive study drug as long as there is clinical benefit and in absence of intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid malignancy that is metastatic or unresectable, and for which standard curative or palliative measures does not exist or are no longer effective
* Performance status (based on the Eastern Cooperative Oncology Group assessments) of <= 2
* Life expectancy > 3 months
* Adequate gastrointestinal absorption status
* Must meet protocol-defined criteria for lab assessments and adequate bone marrow, liver, and kidney function.

Exclusion Criteria:

* Known central nervous system metastases
* Chemotherapy, radiotherapy, immunotherapy within 4 weeks before study drug administration or incomplete recovery from preceding surgery
* Previous participation in a clinical study with histone deacetylase (HDAC) inhibitor or another investigational anticancer agent within 4 weeks of dosing with R306465
* Patient has signs and symptoms of acute infection requiring systemic therapy
* Patient is not recovered from reversible toxicity of prior anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety and maximum tolerated dose of R306465 when given as a daily oral dose during 3 weeks followed by a 1 week recovery period. Study the absorption, break down and elimination of R306465 following oral administration.

SECONDARY OUTCOMES:
Investigate the effect of food on oral administration of R306465. Evaluate the antitumor activity of R306465 in patients with measurable cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.